CLINICAL TRIAL: NCT06928103
Title: Comparison of the Acute Effects of Different Warm-up Protocols on Shoulder Mobility, Muscle Stiffness, Muscle Power Performance, Shoulder Functional Ability and Shoulder Endurance in Overhead Athletes With Posterior Shoulder Tightness
Brief Title: Comparison of the Acute Effects of Different Warm-up Protocols in Overhead Athletes With Posterior Shoulder Tightness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU113009AF
Record Dates: First submitted 2025-03-26; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-09

CONDITIONS: Posterior Shoulder Tightness
Keywords: Posterior Shoulder Tightness
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dynamic stretching group (Active Comparator)
  Interventions: Other: Dynamic stretching
- Static stretching and Dynamic stretching group (Experimental)
  Interventions: Other: Static stretching and dynamic stretching
- Dynamic stretching and foam rolloing group (Experimental)
  Interventions: Other: Dynamic stretching and foam rolling

INTERVENTIONS:
Other: Dynamic stretching — dynamic stretching: teach the participants movements that they can perform to warm up their soft tissues.
  Arms: Dynamic stretching group
Other: Static stretching and dynamic stretching — Static stretching: help patients do the movement that they're limited to stretch their soft tissue; Dynamic stretching: teach the participants movements that they can perform to warm up their soft tissues
  Arms: Static stretching and Dynamic stretching group
Other: Dynamic stretching and foam rolling — Dynamic stretching: teach the participants movements that they can perform to warm up their soft tissues; Foam rolling: Teach the participants how to use a massage ball so that they can perform movements to warm up their soft tissues
  Arms: Dynamic stretching and foam rolloing group

SUMMARY:
The aim of this study is to investigate the immediate effects of different warm-up protocols on Shoulder mobility, Muscle stiffness, Muscle power performance, Shoulder functional ability and Shoulder endurance in overhead athletes with posterior shoulder tightness

ELIGIBILITY:
Inclusion Criteria:

* Recreational or amateur athletes between the ages of 18 and 40
* Training time exceeding four hours per week
* Shoulder internal rotation is reduced by more than 15 degrees compared to the non-dominant side, or the sum of shoulder external rotation and internal rotation is less than 15 degrees compared to the non-dominant side or Shoulder horizontal adduction is reduced by move than 15 degrees compared to the non-dominant side

Exclusion Criteria:

* Shoulder pain within the past three months
* History of shoulder fracture, dislocation, or soft tissue tear surgery in the past
* Contraindications for massage include: open wounds in the treatment area, skin cancer, infections in the treatment area, and severe edema

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-01-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Passive range of motion | Pre-intervention and post intervention (immediate effect)
  Passive range of motion (PROM) testing includes shoulder internal rotation, external rotation, and horizontal adduction.
  For shoulder internal and external rotation, the subject lies supine on a treatment table with the shoulder abducted to 90° and the elbow flexed to 90°. One examiner stabilizes the humeral head while passively moving the arm, and another examiner measures the range using a goniometer.
  For shoulder horizontal adduction, the subject lies supine with the shoulder flexed to 90°, the elbow flexed to 90°, and the shoulder internally rotated. One examiner stabilizes the scapula while passively moving the arm, and another examiner measures the range using a goniometer.
  (unit of measure : degree)
Active range of motion | Pre-intervention and post intervention (immediate effect)
  Active range of motion (AROM) testing includes shoulder internal rotation, external rotation, and horizontal adduction.
  For shoulder internal and external rotation, the subject lies supine on a treatment table with the shoulder abducted to 90° and the elbow flexed to 90°. One examiner stabilizes the humeral head while the subject actively performs the movement, and another examiner measures the range using a goniometer.
  For shoulder horizontal adduction, the subject lies supine with the shoulder flexed to 90°, the elbow flexed to 90°, and the shoulder internally rotated. One examiner stabilizes the scapula while the subject actively performs the movement, and another examiner measures the range using a goniometer.
  (unit of measure : degree)
Muscle stiffness | Pre-intervention and post intervention (immediate effect)
  The stiffness of the posterior shoulder muscles is assessed using a myotonometer (Myoton-Pro, Myoton AS, Tallinn, Estonia) to measure the infraspinatus and posterior deltoid.
  During the test, the subject exposes the shoulder area and lies in a prone position. A towel is placed under the front of the shoulder to ensure relaxation.
  For the infraspinatus, the measurement is taken two finger-widths below the midpoint of the scapular spine. For the posterior deltoid, the measurement is taken two finger-widths from the inferior edge of the acromion. Each muscle is tested five times, and the average value is recorded.
  (unit of measure : Newton metre)
Power performance | Pre-intervention and post intervention (immediate effect)
  Shoulder internal and external rotation strength is assessed with the subject lying supine on a treatment table, with the shoulder abducted to 90° and the elbow flexed to 90°.
  The subject is instructed to perform a maximal isometric contraction of internal or external rotation for 3 seconds at the highest speed and force possible. One examiner stabilizes the humeral head, while a handheld dynamometer (Kinvent, Montpellier, France) attached to a handle is used for measurement.
  The test is performed three times, with a 30-second rest between trials, and the average value is recorded.
  (unit of measure : kilogram and Kilogram Per Second)

SECONDARY OUTCOMES:
Functional performance - Y balance test upper quarter | Pre-intervention and post intervention (immediate effect)
  Before performing the Y Balance Test upper quarter (Move2Perform, Evansville, IN, USA), the subject removes shoes and socks and assumes a push-up position with feet shoulder-width apart.
  The starting position is set with the dominant hand placed on the platform, aligning the adducted thumb with the red line.
  The test involves reaching in three directions-lateral, diagonal-up, and diagonal-down-using the non-dominant hand while returning to the starting position after each reach. Each direction is tested three times, and the average value is recorded.
  (unit of measure : centimetre)
Functional performance - closed kinetic chain upper extremity stability test (CKCUEST) | Pre-intervention and post intervention (immediate effect)
  The Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) measures upper limb dynamic stability and plyometric ability.
  To ensure accuracy, the distance from C7 to the tip of the middle finger is measured to determine hand placement.
  During the test, the subject assumes a push-up position with feet together and alternately touches the opposite hand as many times as possible within 15 seconds. The test is performed twice, with a 45-second rest between trials, and the average value is recorded.
  (unit of measure : times)
Shoulder endurance | Pre-intervention and post intervention (immediate effect)
  The Posterior Shoulder Endurance Test assesses the fatigue resistance of posterior shoulder muscles.
  Before testing, a standardized dumbbell weight is determined as 2% of the subject's body weight, rounded to the nearest value.
  The subject lies prone at the edge of a treatment table with the head turned toward the testing side and the arm hanging naturally.
  Following a 60 Hz rhythm, the subject repeatedly lifts the arm sideways (shoulder external rotation, 90° horizontal abduction, and full elbow extension) until unable to continue or compensatory movements occur.
  (unit of measure : times)

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Yang Ming Chiao Tung University, Taipei
  - No. 155, Sec. 2, Linong St. Beitou Dist., Taipei City 112304, Taiwan, Taipei